CLINICAL TRIAL: NCT05609630
Title: A Multicenter, Randomized Open-Label Study to Assess the Efficacy, Safety, and Pharmacokinetics of Upadacitinib With a Tocilizumab Reference Arm in Subjects From 1 Year to Less Than 18 Years Old With Active Systemic Juvenile Idiopathic Arthritis
Brief Title: Study of Oral Upadacitinib and Subcutaneous/Intravenous Tocilizumab to Evaluate Change in Disease Activity, Adverse Events and How Drug Moves Through the Body of Pediatric and Adolescent Participants With Active Systemic Juvenile Idiopathic Arthritis.
Acronym: SELECT-sJIA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-682; 2022-501599-25-00 (Other: EU CT)
Record Dates: First submitted 2022-11-07; First posted 2022-11-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Systemic Juvenile Idiopathic Arthritis; sJIA; Upadacitinib; ABT-494
MeSH Terms: conditions — Arthritis, Juvenile | interventions — upadacitinib; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1 Upadacitinib (Experimental): Participants will receive upadacitinib for 52 weeks.
  Interventions: Drug: Upadacitinib
- Cohort 1 Tocilizumab (Active Comparator): Participants will receive tocilizumab for 52 weeks.
  Interventions: Drug: Tocilizumab
- Cohort 2 Upadacitinib (Experimental): Participants will receive upadacitinib for 52 weeks.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Oral tablet or Oral solution
  Other Names: RINVOQ; ABT-494
  Arms: Cohort 1 Upadacitinib; Cohort 2 Upadacitinib
Drug: Tocilizumab — Subcutaneous injection or Intravenous infusion
  Arms: Cohort 1 Tocilizumab

SUMMARY:
Juvenile Idiopathic Arthritis (JIA) is the most common type of arthritis that affects children. The term "idiopathic" means "of unknown origin". It is a chronic (long-lasting) disease that causes swelling, warmth, and pain of one or more small joints. Systemic JIA ia a rare and serious form of JIA. Systemic" means it may affect not only the joints but other parts of the body, including the liver, lungs and heart. sJIA is more severe and can be more challenging to diagnose and treat than other types of juvenile idiopathic arthritis. It is a lifelong disease for many patients and can continue into adulthood. This study will assess how safe and effective upadacitinib is in treating pediatric and adolescent participants aged 1 to < 18 with systemic juvenile idiopathic arthritis (sJIA) and will include a tocilizumab treatment arm for reference. Adverse events and change in the disease activity will be assessed.

Upadacitinib is an investigational drug being developed for the treatment of sJIA. Participants are assigned to 1 of 2 cohorts. In cohort 1, participants will receive upadacitinib or tocilizumab reference. In cohort 2, participants will receive upadacitinib. Approximately 90 participants with sJIA will be enrolled in approximately 45 sites worldwide.

Participants will receive upadacitinib oral tablets once daily or oral solution twice daily or tocilizumab subcutaneous injection or intravenous infusion as per local label for 52 weeks and followed for approximately 30 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits/calls during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- Baseline with a total body weight of 10 kg or higher at screening and symptoms of systemic juvenile idiopathic arthritis (sJIA) according to International League of Associations for Rheumatology (ILAR) criteria for at least 6 weeks prior to Screening, with onset prior to 16 years old, and meet the following conditions:

* Must have active sJIA with at least 2 active joints at Screening and Baseline, fever more than 38°C on at least one day within 14 consecutive days before the Screening Visit, and an erythrocyte sedimentation rate (ESR) or high-sensitivity C-reactive protein (hsCRP) > upper limit of normal (ULN) at Screening. OR At least 4 active joints at Screening and Baseline and an ESR or hsCRP > ULN at Screening.
* Must have inadequate response to previous treatment with nonsteroidal anti-inflammatory drugs and/or systemic glucocorticoids, as judged by the investigator.
* For Cohort 1, participants must not have had previous treatment with any IL-6 inhibitor. For Cohort 2, participants must have an intolerance or inadequate response to an IL-6 inhibitor as judged by the investigator.

Note: For Cohort 1, participants must be ages 2 to < 18 years old in countries where SC tocilizumab is not approved for sJIA.

Exclusion Criteria:

* Has any type of juvenile idiopathic arthritis (JIA), other than sJIA, as defined by the ILAR criteria, and must not have a history or presence of any other autoimmune inflammatory condition other than sJIA.
* Has uncontrolled severe systemic disease and/or impeding or active macrophage activation syndrome within 1 month prior to Baseline.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Adapted systemic Juvenile Idiopathic Arthritis (sJIA) American College of Rheumatology (ACR) 30 Response | At Week 12
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant. ACR 30 Response is defined as absence of fever [> 38°C] in the previous 1 week preceding evaluation and improvement of ≥ 30% of the 6 variables of the JIA core set with no more than 1 variable worsening by > 30%.
Number of Participants with Adverse Events (AEs) | Up to Approximately Week 52
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Adapted systemic Juvenile Idiopathic Arthritis (sJIA) American College of Rheumatology (ACR) 50 Response | Week 12
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant. ACR 50 Response is defined as absence of fever [> 38°C] in the previous 1 week preceding evaluation and improvement of ≥ 50% of the 6 variables of the JIA core set.
Percentage of Participants Achieving Adapted systemic Juvenile Idiopathic Arthritis (sJIA) American College of Rheumatology (ACR) 70 Response | Week 12
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant. ACR 70 Response is defined as absence of fever [> 38°C] in the previous 1 week preceding evaluation and improvement of ≥ 70% of the 6 variables of the JIA core set.
Percentage of Participants Achieving Adapted systemic Juvenile Idiopathic Arthritis (sJIA) American College of Rheumatology (ACR) 90 Response | Week 12
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant. ACR 90 Response is defined as absence of fever [> 38°C] in the previous 1 week preceding evaluation and improvement of ≥ 90% of the 6 variables of the JIA core set.
Percentage of Participants Achieving Adapted systemic Juvenile Idiopathic Arthritis (sJIA) American College of Rheumatology (ACR) 100 Response | Week 12
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant. ACR 100 Response is defined as absence of fever [> 38°C] in the previous 1 week preceding evaluation and improvement of ≥ 100% of the 6 variables of the JIA core set.
Change from Baseline in Number of Joints with Active Arthritis | Week 12
  Change from Baseline in Number of Joints with Active Arthritis
Change from Baseline in Number of Joints with Limitation of Motion | Week 12
  Change from Baseline in Number of Joints with Limitation of Motion
Change from Baseline in Childhood Health Assessment Questionnaire-Disability Index (CHAQ-DI) | Week 12
  The CHAQ-DI consists of 30 items and assesses function in 8 areas: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities. There are 5 response options ranging from no difficulty to unable to do, scored 0 to 3, and not applicable.
Change From Baseline in Patient's Global Assessment (PtGA) | Week 12
  Participants rated their disease activity for the past 24 hours using a Patient's Global Assessment of Disease Activity Global visual analogue scale (VAS). The range is 0 to 100 mm, with 0 representing no disease activity and 100 representing severe disease activity. Negative values indicate improvement from baseline.
Change From Baseline in Physician's Global Assessment of Disease Activity (PhGA) | Week 12
  Participants rated their disease activity for the past 24 hours using a Patient's Global Assessment of Disease Activity Global visual analogue scale (VAS). The range is 0 to 100 mm, with 0 representing no disease activity and 100 representing severe disease activity. Negative values indicate improvement from baseline.
Change From Baseline in High-Sensitivity C-Reactive Protein (hsCRP) | Week 12
  High sensitivity C-reactive protein was analyzed by a central laboratory. The median percent change from baseline in CRP is assessed at each time point.
Percentage of Participants with Absence of fever (> 38°C) Attributed to systemic Juvenile Idiopathic Arthritis (sJIA) | Week 12
  Absence of fever (> 38°C) Attributed to systemic Juvenile Idiopathic Arthritis (sJIA)
Change from Baseline in Glucocorticoid Dose | Week 12
  Change from Baseline in Glucocorticoid Dose
Change from Baseline in Juvenile Arthritis Disease Activity Score (JADAS27-CRP) | Week 12
  Juvenile Arthritis Disease Activity Score (JADAS27-CRP) will be assessed
Percentage of Participants Achieving Inactive Disease (ID) Status by Juvenile Arthritis Disease Activity Score (JADAS27)-CRP | Week 12
  Inactive Disease (ID) status by 27-joint Juvenile Arthritis Disease Activity Score (JADAS27)-CRP will be assessed.
Percentage of Participants Achieving Minimal Disease Activity (MDA) by Juvenile Arthritis Disease Activity Score (JADAS27)-CRP | Week 12
  Minimal Disease Activity (MDA) by 27-joint Juvenile Arthritis Disease Activity Score (JADAS27)-CRP will be assessed.
Percentage of Participants Achieving Clinical Remission by Juvenile Arthritis Disease Activity Score (JADAS27)-CRP | Week 12
  Clinical Remission by 27-joint Juvenile Arthritis Disease Activity Score (JADAS27)-CRP will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (44):
- United States (6):
  - Phoenix Children's Hospital /ID# 253403, Phoenix, Arizona
  - Childrens National Medical Center /ID# 253344, Washington D.C., District of Columbia
  - New York Medical College /ID# 253437, Valhalla, New York
  - Levine Children's Hospital /ID# 253491, Charlotte, North Carolina
  - Cincinnati Childrens Hospital Medical Center /ID# 251827, Cincinnati, Ohio
  - Randall Children's Hospital /ID# 251829, Portland, Oregon
- Argentina (3):
  - Instituto CAICI S.R.L /ID# 251448, Rosario, Santa Fe Province
  - Centro de Investigaciones Medicas Tucuman /ID# 251781, San Miguel de Tucumán, Tucumán Province
  - Hospital de Niños de la Santisima Trinidad /ID# 252736, Córdoba
- Australia (2):
  - Monash Health - Monash Medical Centre /ID# 251691, Clayton, Victoria
  - Royal Children's Hospital /ID# 251663, Parkville, Victoria
- Landeskrankenhaus Bregenz /ID# 266317, Bregenz, Vorarlberg, Austria
- Brazil (3):
  - CMiP - Centro Mineiro de Pesquisa Ltda - ME /ID# 251769, Juiz de Fora, Minas Gerais
  - Hospital Sao Paulo /ID# 251765, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 251764, São Paulo
- China (5):
  - The Childrens Hospital of Chongqing Medical University /ID# 251539, Chongqing, Chongqing Municipality
  - Children'S Hospital Of Soochow University /ID# 251755, Suzhou, Jiangsu
  - Xi'an Children's Hospital /ID# 251693, Xi'an, Shaanxi
  - Children's Hospital of Fudan University /ID# 251619, Shanghai, Shanghai Municipality
  - The Children's Hospital of Zhejiang University School of Medicine /ID# 251754, Hangzhou, Zhejiang
- Germany (4):
  - Universitaetsklinikum Freiburg /ID# 253288, Freiburg im Breisgau, Baden-Wurttemberg
  - Asklepios Klinik Sankt Augustin /ID# 251565, Sankt Augustin, North Rhine-Westphalia
  - St. Josef-Stift Sendenhorst /ID# 268680, Sendenhorst, North Rhine-Westphalia
  - Hamburger Zentrum fuer Kinder- und Jugendrheumatologie /ID# 251564, Hamburg
- Semmelweis Egyetem /ID# 266750, Budapest, Hungary
- Italy (2):
  - Azienda Ospedaliero Universitaria Meyer /ID# 251775, Florence, Firenze
  - IRCCS Istituto Giannina Gaslini /ID# 251776, Genoa, Genova
- Japan (5):
  - Hyogo Prefectural Kobe Children'S Hospital - Minatojima /ID# 251649, Kobe, Hyōgo
  - St Marianna University School Of Medicine /ID# 251623, Kawasaki-shi, Kanagawa
  - Niigata University Medical & Dental Hospital /ID# 251538, Niigata, Niigata
  - Osaka Medical and Pharmaceutical University Hospital /ID# 252092, Takatsuki-shi, Osaka
  - Institute of Science Tokyo Hospital /ID# 251505, Bunkyo-ku, Tokyo
- CREA de Guadalajara SC /ID# 252917, Guadalajara, Jalisco, Mexico
- Universitair Medisch Centrum Utrecht /ID# 267435, Utrecht, Netherlands
- Spain (2):
  - Hospital Sant Joan de Deu /ID# 251353, Esplugues de Llobregat, Barcelona
  - Hospital Universitario y Politecnico La Fe /ID# 251352, Valencia
- Queen Silvia Children's Hosp /ID# 251318, Gothenburg, Västra Götaland County, Sweden
- Taiwan (2):
  - National Taiwan University Hospital /ID# 267387, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 267390, Taoyuan
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty /ID# 253677, Ankara
  - Istanbul University Istanbul Medical Faculty /ID# 251652, Istanbul
  - Istanbul Universitesi-Cerrahpasa Cerrahpasa Tip Fakultesi /ID# 251651, Istanbul
  - Umraniye Training and Res Hosp /ID# 251653, Istanbul
- Great Ormond Street Children's Hospital /ID# 251512, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related info — https://www.abbvieclinicaltrials.com/study/?id=M14-682